CLINICAL TRIAL: NCT04127149
Title: Pragmatic Evaluation of Ultra-portable Ultrasound for a List of Indications in General Practice
Brief Title: Evaluation of Ultra-portable Ultrasound in General Practice
Acronym: EPEMedG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL18_1004
Record Dates: First submitted 2019-10-08; First posted 2019-10-15 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Pneumonia; Pleural Effusion; Renal Colic; Hepatic Colic or Cholecystitis; Subcutaneous Abscess or Cyst; Fracture of Long Bones; Intra-uterine Pregnancy or Extra-uterine Pregnancy or Miscarriage; Phlebitis
Keywords: ultrasound scanner; sonogram; general practice
MeSH Terms: conditions — Pneumonia; Pleural Effusion; Renal Colic; Cholecystitis; Cysts; Pregnancy, Ectopic; Abortion, Spontaneous; Phlebitis | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group with ultrasound (Experimental): The first group consists of nine general practitioners having received a brief training on the use of ultrasound scanners in general practice. The general practitioner includes all adult patients who are consulting for one of the 8 medical conditions studied and perform an ultrasound scan. Two weeks later, he/she calls each patient to collect the necessary data.
  Interventions: Diagnostic Test: Ultrasound scan
- Group without ultrasound (No Intervention): The second group consists of nine general practitioners. Each physician includes all adult patients who are consulting for one of the 8 medical conditions studied and performs a standard consultation. Two weeks later, he/she calls each patient to collect the necessary data.

INTERVENTIONS:
Diagnostic Test: Ultrasound scan — The group uses an ultrasound device for the consultation.
  Arms: Group with ultrasound

SUMMARY:
This is an interventional multi-centre study comparing two groups of general practitioners with or without an ultrasound scanner over a period of 6 months. The evaluation focuses on the management of patients for 8 pathologies:

* Pneumonia
* Pleural effusion
* Renal colic
* Hepatic colic or cholecystitis
* Subcutaneous abscess or cyst
* Fracture of long bones
* Intra-uterine pregnancy or extra-uterine pregnancy or miscarriage
* Phlebitis The principal hypothesis is that there are fewer complementary exams in the group of doctors using ultrasound scanners.

The secondary hypotheses are:

* There is better patient orientation (emergency care, specialist consultation, return home) in the group of doctors using the ultrasound scanners.
* The global cost of the care is lower in the group of doctors using the ultrasound.
* Using ultrasound during the consultation decreases the anxiety of the patient.
* Using ultrasound increases the duration of the consultation.
* There is no difference between the predicted and the real orientation of the patients.

ELIGIBILITY:
Inclusion Criteria:

* patients age 18 and over
* consulting their general practitioner for one of the 8 conditions below

Exclusion Criteria:

* patients who have already received an imagery exam for the acute episode justifying the consult
* opposition to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-10-20 (Actual)

PRIMARY OUTCOMES:
Number of complementary exams | Two weeks after inclusion
  Two weeks after the initial consultation, with or without ultrasound scanners, the general practitioners call their patients to know:
  * The number of imagery exams they had (ultrasound, MRI, scanner, radiology…)
  * The number of biological analysis (CRP, ASAT, ALAT, Lipase…)

SECONDARY OUTCOMES:
Number of hospitalisations, specialist orientation or return home | Two weeks after inclusion
  Two weeks after the initial consultation, with or without ultrasound scanners, the general practitioners call their patients to know if within the past two weeks, they have been hospitalised, required emergency care, needed to consult a specialist, or returned back home
Cost of care | Four weeks after inclusion in the study
  After knowing the patient orientation and the complementary exams they had, an estimation of the cost of care is made.
Anxiety score measured by the State-Trait Anxiety Inventory (STAI-Y) scale | Two weeks after inclusion in the study
  Two weeks after the initial consultation, with or without ultrasound scanners, the general practitioners call their patients to know the result of the anxiety test they took the day of the first consultation.
Consultation duration | Two weeks after inclusion in the study
  The day of the first consultation, the general practitioner writes the time spent

CONTACTS AND LOCATIONS:
Overall Officials: Francis PELLET, MD, Principal Investigator — Maison de sante pluridisciplinaire Leopold Ollier Les Vans
Locations (1):
- Maison de santé pluridisciplinaire Léopold Ollier, Les Vans, France

REFERENCES:
- [Result] Dasse-Hartaut J, Couture S. Pragmatic evaluation of handheld point-of-care ultrasound in general practice. MD thesis. Claude Bernard University Lyon 1; 2021. Thesis supervisor: Dr Francis Pellet.